CLINICAL TRIAL: NCT04511988
Title: Evaluation of Clonal Heterogeneity and Tumor Evolution Using Liquid Biopsy in Newly Diagnosed Patients With High Grade Adenocarcinoma of Ovarian Origin, Fallopian Tubes or Primary Peritoneal
Brief Title: Using Liquid Biopsy in Newly Diagnosed Patients With High Grade Adenocarcinoma of Ovarian Origin, Fallopian Tubes or Primary Peritoneal
Acronym: BOVARY CE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02251-38
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): blood sample (20 ml) and biopsy
  Interventions: Other: Diagnostic Test

INTERVENTIONS:
Other: Diagnostic Test — blood sample (20 ml) and biopsy

SUMMARY:
BOVARY-CE is a monocentric, pilot, longitudinal, real-life study with a total duration of 36 months. The purpose of this study is to assess the feasibility of using liquid biopsy as a substitute for tissue multisampling, in order to describe clonal heterogeneity and tumor evolution in patients with ovarian cancer. The method involves the inclusion of 20 patients with high-grade ovarian adenocarcinoma, fallopian tubes or primary peritoneal origin, not pretreated, newly diagnosed, and eligible for treatment who will participate in the research. These patients will have several samples throughout their treatment for a period of 2 years: blood samples which will be taken at each therapeutic moment of interest.

Tissue samples which will be taken at the time of the diagnostic laparoscopy and at the time of surgery.

The concentration of cfDNA and tumor heterogeneity will be used to predict disease-related events defined as relapse, progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with non-treated high grade serous and endometrioid carcinoma of ovarian, fallopian tube, or primary peritoneal origin proven cytologically or histologically at inclusion and eligible for treatment
* Patient eligible for an upfront surgery or pretherapeutic coelioscopy
* Adequate haemoglobin rate ≥ 9 g/dL
* Patient affiliated to a social security scheme
* Ability to provide written informed consent

Exclusion Criteria:

* Age < 18 years
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Contraindication to blood samples of 20 mL
* Pregnant or breast-feeding women
* Ongoing treatment for the newly diagnosed cancer or the recurrence
* Other cancers treated within the last 5 years
* Patient under guardianship or curatorship or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Using the concentration of cfDNA to predict disease events | 12 months
  cfDNA concentration (ng / µl)

CONTACTS AND LOCATIONS:
Overall Officials: LEUFFLEN Léa, MD PhD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided